CLINICAL TRIAL: NCT01173965
Title: Treatment of Dysfunctional Uterine Bleeding With Second Generation Ablation Devices: Microwaves (MEA®) vs Bipolar Impedance Control System (Novasure®)
Brief Title: Endometrial Ablation With Non-hysteroscopic Methods
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: George Pados, 1st Dept Of ObGyn, "Papageorgiou" General Hospital, Medical School, Aristotle University of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3873
Record Dates: First submitted 2010-08-02; First posted 2010-08-03 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2009-09

CONDITIONS: Dysfunctional Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endometrial ablation with microwaves (Active Comparator): Endometrial ablation with the use of MEA(microwaves endometrial ablation device)
  Interventions: Device: MEA
- Endometrial ablation with bipolar diathermy (Active Comparator): Endometrial ablation with Novasure(bipolar impedence control system)
  Interventions: Device: Novasure

INTERVENTIONS:
Device: MEA — Microwave endometrial ablation device
  Other Names: Microwaves (MEA®)
  Arms: Endometrial ablation with microwaves
Device: Novasure — Bipolar impedence control system
  Other Names: Bipolar Impedance Control System (Novasure®)
  Arms: Endometrial ablation with bipolar diathermy

SUMMARY:
Endometrial ablation in women with dysfunctional uterine bleeding using second generation ablation devices is a common widespread therapeutic approach. This study aims to prove that amenorrhoea rates using Novasure are higher than those observed in microwave endometrial ablation, one year following intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting with dysfunctional uterine bleeding having completed their family planning(no wish for further childbearing)

Exclusion Criteria:

* Endometrial pathology
* FSH > 20 day 2 -day 3 of the cycle
* Clotting Disorders
* Thyroid Dysfunction

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2008-01; Primary Completion 2010-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Amenorrhoea rates one year after intervention

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - First Dept. Of ObGyn, Medical School Aristotle University of Thessaloniki, Papageorgiou Hospital, Thessaloniki, Thessaloniki
  - First Dept. of ObGyn, Medical School, Aristotle University of Thessaloniki, Papageorgiou Hospital, Thessaloniki, Thessaloniki